CLINICAL TRIAL: NCT05738863
Title: The Effect of Repetative Transcranial Magnetic Stimulation Therapy on Lower Urinary System Dysfunctions in Stroke Patients
Brief Title: The Effect of Repetative Transcranial Magnetic Stimulation Therapy for Stroke Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Afyonkarahisar Health Sciences University (Other)
Responsible Party: Principal Investigator, Ayşenur Beysel, Research Assistant Doctor, Afyonkarahisar Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 586
Record Dates: First submitted 2023-02-13; First posted 2023-02-22 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Lower Urinary Tract Symptoms
Keywords: hemiplegia; urinary dysfunction; detrusor overactivity
MeSH Terms: conditions — Lower Urinary Tract Symptoms; Hemiplegia; Urinary Bladder, Overactive

STUDY DESIGN:
Intervention Model Description: Effects of Repetative Transcranial Magnetic Stimulation Therapy on Lower Urinary System Dysfunctions in Stroke Patients; A Randomized Study of Double Blind With Sham Control
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Frequency rTMS Protocol (Experimental): It was planned to apply 1 Hz low-frequency inhibition protocol to the primary motor cortex 5 days a week for 3 weeks, for a total of 15 sessions.
  Interventions: Device: Low Frequency rTMS Protocol
- Sham rTMS Protocol (Placebo Comparator): It was planned to apply the recorded beat sound to the primary motor cortex area daily 5 days a week for 3 weeks, for a total of 15 sessions by turning the TMS coil with the reverse side and in a 90-angle upright position.
  Interventions: Device: Sham rTMS Protocol

INTERVENTIONS:
Device: Low Frequency rTMS Protocol — It was planned to apply 1 Hz low-frequency inhibition protocol to the primary motor cortex 5 days a week for 3 weeks, for a total of 15 sessions.
  rTMS application Magventure MagPro R30 device is planned to provide magnetic stimulation with its stimulator. The stimulation pattern was shaped according to the protocols used in previous studies.
  All patients were planned to continue the neurological rehabilitation program throughout the study.
  Along with the daily rTMS session, patients will continue to use the drugs in the medical treatment they are using and the drugs started for incontinence at the same effective dose, and no new incontinence medication will be started and the dose will not be changed during the rTMS sessions.
  Arms: Low Frequency rTMS Protocol
Device: Sham rTMS Protocol — It was planned to apply the recorded beat sound to the primary motor cortex area daily 5 days a week for 3 weeks, for a total of 15 sessions by turning the TMS coil with the reverse side and in a 90-angle upright position.
  All patients were planned to continue the neurological rehabilitation program throughout the study.
  Along with the daily rTMS session, patients will continue to use the drugs in the medical treatment they are using and the drugs started for incontinence at the same effective dose, and no new incontinence medication will be started and the dose will not be changed during the rTMS sessions.
  Arms: Sham rTMS Protocol

SUMMARY:
The aim of our study is to investigate the effect of repetitive transcranial magnetic stimulation therapy (rTMS) on lower urinary system dysfunctions and detrusor muscle activity in stroke patients.

DETAILED DESCRIPTION:
Stroke is the second leading cause of death in adults and one of the major causes of long-term disability. Functional limitations that develop in the post-stroke period affect the quality of life and activities of daily living of the patients. The main purpose of stroke rehabilitation is to improve the quality of life of patients in the areas of physical, functional, psychological and social health.

Post-stroke urinary incontinence (PSUI) is a common complication that manifests as involuntary loss of urine. It has been reported that post-stroke urinary incontinence (PSUI) affects 40-60% of patients admitted to the hospital after stroke, up to 25% still have problems when they are discharged from the hospital, and 15% remain incontinence one year later. Recent studies have shown that 79% of stroke survivors develop urinary incontinence.

It has been reported that this complication is also associated with psychological problems such as low self-esteem and anxiety. In addition, the presence of urinary incontinence has been considered a marker of stroke severity and a higher mortality rate than those without urinary incontinence. Therefore, Post-stroke urinary incontinence (PSUI) management is critical and should be the goal of all stroke health professionals.

In recent years, there is a need for more effective approaches on neuroplasticity mechanisms in stroke rehabilitation. Repetitive transcranial magnetic stimulation (rTMS) is an innovative approach applied in this field. With the application of repetitive transcranial magnetic stimulation (rTMS), it is aimed to modulate plasticity and restore the normal activity pattern.

Repetitive transcranial magnetic stimulation (rTMS) is a painless non-invasive technique widely used in clinical routine practice to modulate the neural excitability of the human brain. High frequency rTMS (>5 Hz) increases neural activity (long term potentiation), while low frequency (1 Hz) rTMS decreases neural activity (long term depression).

Previous studies have shown that detrusor overactivity (DO) constitutes the major urodynamic model of post-stroke urinary incontinence (PSUI).This suggests that the brain, which is the center of incontinence with detrusor overactivity, is a potential target for therapeutic interventions.

Repetitive transcranial magnetic stimulation (rTMS) is a newly developed noninvasive brain stimulation method for the treatment of neurological disorders.When applied to cortical areas corresponding to the pelvic region, it can modulate cortical excitability and induce long-lasting neuroplastic changes.

High-frequency rTMS (>5 Hz) increases neural activity (long-term potentiation), low-frequency (1 Hz) rTMS decreases neural activity. (long-term depression). Clinical studies have shown that inhibition of bladder activity is possible with low frequency (≤ 1 Hz) rTMS in the primary motor cortex (M1).

Our primary aim is to investigate the effect of low-frequency rTMS treatment on urinary system dysfunctions in the primary motor cortex (M1) in stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* A person between the ages of 40-80 who applied to AFSU Physical Medicine and Rehabilitation Clinic with the diagnosis of stroke in the inpatient service or outpatient for neurological rehabilitation,
* Having had a stroke at least three months ago,
* Able to follow two-stage verbal commands and agree to participate in the study voluntarily and regularly,
* Medically stable,
* Neurologically stable,
* After taking the anamnesis and physical examination, patients who meet the inclusion criteria and whose exclusion criteria were excluded will be included in the study

Exclusion Criteria:

* Patients with significant comorbidities such as severe heart disease (aortic stenosis, angina, hypertrophic cardiomyopathy, arrhythmia, pacemaker) and uncontrolled hypertension,
* Epilepsy, history of antiepileptic drug use intracranial metal body,
* Having an ear implant,
* Cognitive dysfunction,
* Lower extremity peripheral nerve injury
* Malignancy
* Active infection
* Infection on the skin in the application area, open wound
* İnflammatory disease
* Orthopedic injuries that can limit maximal effort contractions
* Brain lesion or history of drug use that may affect seizure threshold
* İncreased intracranial pressure
* Patients with uncontrolled migraine

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2022-12-02 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Danish Scale at 15th day and 8th week | up to 8th week
  The questionnaire consists of 12 questions about lower urinary tract symptoms (LUTS). It is a questionnaire study that questions the frequency and severity of their symptoms (symptom score) and its effect on their daily life (discomfort score) from the participants. It is one of the reliable methods that questions the frequency and severity of lower urinary tract symptoms and disturbing factors.
Change from baseline International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form (ICIQ-UI SF) at 15th day and 8th week | up to 8th week
  Evaluates the severity of urinary incontinence symptoms and their impact on health-related quality of life. When using the ICIQ-UI SF, an overall ICIQ score in the range of 0-21 is obtained from the first three questions. A score of zero means no urine leakage and no impact on quality of life. Question 1 (Q1) measures the frequency of urinary incontinence, question 2 (Q2) evaluates the amount of leakage, and question 3 (Q3) evaluates how much urinary incontinence affects daily life.

SECONDARY OUTCOMES:
Change from baseline Uroflowmetry and residual urine at 15th day and 8th week | up to 8th week
  It is one of the ideal follow-up methods due to its ease and non-invasiveness in the evaluation of lower urinary system dysfunction. The maximum flow rate, mean flow rate, voided volume, and the corresponding postvoid residual urine are evaluated.
Change from baseline Overactive Bladder Symptom Score (OABSS) at 15th day and 8th week | up to 8th week
  It includes questions that address the four symptoms of overactive bladder (daytime frequency, nighttime frequency, urgency, urge to incontinence) designed to measure overactive bladder symptoms as a single score. It is a test consisting of questions such as how many times the need to urinate after waking up in the morning before going to sleep, how many times the need to wake up to urinate from sleep to wake up in the morning, how often the urge to urinate is difficult to postpone, and how often urine is leaked because the sudden urge to urinate cannot be delayed.
Change from baseline Urinary Incontinence Quality Of Life Scale at 15th day and 8th week | up to 8th week
  It has been shown to be useful in clinical practice to evaluate the effects of lower urinary system dysfunction on individuals, the discomfort, embarrassment, withdrawal from social life and deterioration in interpersonal relationships on individual lives; It is an assessment consisting of 22 questions that can cover different areas and characterize symptom severity as well as deterioration in lifestyle.
Change from baseline Barthel İndex at 15th day and 8th week | up to 8th week
  It is a measure of independence in activities of daily living. It is a daily life activity index consisting of 10 questions consisting of nutrition, transfer from wheelchair, self-care, sitting on the toilet, bathing, walking on the right floor, using a wheelchair, going up and down stairs, dressing, undressing, bowel care, bladder care.
Change from baseline Beck's Depression Inventory at 15th day and 8th week | up to 8th week
  t is a self-assessment scale that can be used in healthy patient groups to determine the risk of depression in the individual and to measure the level and severity of depressive symptoms. It includes a total of 21 self-assessment questions.
  It provides a four-point Likert-type measurement. Each item gets progressively increasing points between 0 and 3, and the total score is obtained by summing them up. The total score ranges from 0 to 63
Change from baseline Quality of Life (Short Form 36 (SF-36)) at 15th day and 8th week [ | up to 8th week
  This is a self-administered scale, which is widely used to measure the quality of life. It was developed to measure the quality of life in patients who have physical illnesses; however, it can also be successfully used in healthy individuals and patients who have psychiatric diseases. SF-36 includes 36 items and surveys eight domains of health, such as physical functionality, physical role limitations, pain, general health, vitality, social functionality, emotional role limitations, and mental health. Total score was between 0 ( disability) and 100 (no disability). Every subgroup of the questionnaire has a score scale between 0 and 100. Every increase in the subgroup of SF-36 questionnaire, which is a positive scoring system, indicates increase in quality of life related to health.

CONTACTS AND LOCATIONS:
Locations (1):
- Afyonkarahisar Health Sciences University, Afyonkarahisar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jiang W, Tang W, Song Y, Feng Y, Zhou Y, Li L, Tan B. Effectiveness of repetitive transcranial magnetic stimulation against poststroke urinary incontinence: a study protocol for a randomized controlled trial. Trials. 2022 Aug 13;23(1):650. doi: 10.1186/s13063-022-06535-y. PMID 35964135
- [Result] Nardone R, Versace V, Sebastianelli L, Brigo F, Golaszewski S, Christova M, Saltuari L, Trinka E. Transcranial magnetic stimulation and bladder function: A systematic review. Clin Neurophysiol. 2019 Nov;130(11):2032-2037. doi: 10.1016/j.clinph.2019.08.020. Epub 2019 Sep 3. PMID 31541980